CLINICAL TRIAL: NCT06529978
Title: Endocardial Mapping with the CoreMap Electrophysiology Mapping System for Persistent Atrial Fibrillation Protocol
Brief Title: Endocardial Mapping with the CoreMap EP Mapping System
Acronym: INvENI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CoreMap Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CD001
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Phase 1- Mapping Only (Experimental): For Phase 1, the goal is to collect and analyze high fidelity endocardial EGMs in patients with persistent and long-standing persistent AF.
  Interventions: Device: CoreMap EP Mapping System Mapping
- Phase 2- Map Guided Ablation (Experimental): The Phase 2 goal is the initial development and evaluation of a CoreMap-guided tailored ablation strategy and to demonstrate safety and chronic efficacy of the CoreMap EP Mapping System.
  Interventions: Device: CoreMap EP Mapping System Mapping; Device: CoreMap EP Mapping System Map-Guided Ablation
- Phase 3 - Map Guided Ablation (Experimental): For Phase 3, the goal is the evaluation of a CoreMap guided tailored ablation strategy and to demonstrate chronic safety and effectiveness in de novo PerAF patients with the CoreMap EP Mapping System.
  Interventions: Device: CoreMap EP Mapping System Mapping; Device: CoreMap EP Mapping System Map-Guided Ablation

INTERVENTIONS:
Device: CoreMap EP Mapping System Mapping — Endocardial mapping to collect and analyze high fidelity endocardial EGMs in patients with persistent and long-standing persistent AF.
Device: CoreMap EP Mapping System Map-Guided Ablation — Initial development and evaluation of a map-guided tailored ablation strategy and to demonstrate safety and chronic efficacy of the CoreMap EP Mapping System.
  Arms: Phase 2- Map Guided Ablation; Phase 3 - Map Guided Ablation

SUMMARY:
This is a global, multi-site, prospective, feasibility study.

DETAILED DESCRIPTION:
The INvENI Study consists of three phases. For Phase 1, the goal is to collect and analyze high fidelity endocardial electrograms (EGMs) in patients with persistent and long-standing persistent AF. For Phase 2, the goal is the initial development and evaluation of a CoreMap-guided tailored ablation strategy and to demonstrate safety and chronic efficacy of the CoreMap EP Mapping System. For Phase 3, the goal is the evaluation of a CoreMap-guided tailored ablation strategy and to demonstrate both chronic safety and effectiveness in de novo PerAF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has persistent or long-standing persistent AF, at the discretion of the investigator
2. Subject is 18 to 80 years of age
3. Patient scheduled for standard of care AF ablation
4. Subject is able to provide written informed consent
5. Subject is able and willing to complete all study procedures

Exclusion Criteria:

1. Any of the following within three months of enrollment:

   1. Myocardial infarction (MI)
   2. Any surgical or percutaneous cardiac procedure including coronary intervention and cardiac ablation
   3. Confirmed thrombus on imaging
2. Any of the following within six months of enrollment: a) Cardiac surgery including coronary artery bypass grafting, ventriculotomy, atriotomy b) Thromboembolic event (stroke)
3. Any of the following cardiac conditions:

   1. New York Heart Association (NYHA) IV
   2. Left ventricular ejection fraction (LVEF) < 30%
   3. Carotid stenting or endarterectomy
   4. Atrial or ventricular septal closure or left atrial appendage closure
   5. Implanted permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator
   6. Presence of intramural thrombus, tumor (including atrial myxoma), or other abnormality that precludes vascular access, catheter introduction, or manipulation
   7. Unstable angina
   8. Prior mitral or tricuspid valve surgery, repair, prosthetic or mechanical valve
   9. Moderate to severe mitral valve stenosis or other severe valvular disease
   10. Any blood clotting or bleeding abnormalities
4. Contraindication to systemic anticoagulation
5. AF secondary to electrolyte imbalance, acute alcohol intoxication, or reversible or non-cardiac cause
6. Body mass index (BMI) > 40 kg/m2
7. Severe pulmonary disease, pulmonary hypertension, or any chronic respiratory condition
8. Renal failure requiring dialysis or transplant
9. Acute illness, active systemic infection, or sepsis
10. Active drug or alcohol dependency
11. Any contra-indication that may extend procedure time, at the discretion of the operator
12. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence
13. Subject considered part of vulnerable population
14. Life expectancy less than one year
15. Employee of the study site or Sponsor
16. Subjects who are currently enrolled in another study that would directly interfere with this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phases 1 and Phase 2 Primary Endpoint: | 7 days
  Incidence of study device related serious adverse events within seven (7) days of the study procedure.
Phase 2 and Phase 3 Primary Effectiveness Endpoint: | 6 and 12 months
  Chronic Efficacy: Freedom from documented recurrence of AF, lasting longer than 30 seconds (excluding the 90-day blanking period) evaluated at 6 and 12 months.

SECONDARY OUTCOMES:
Phase 1 Secondary Endpoint: | perioperatively/periprocedurally
  Successful completion of the intended study mapping procedure with the CoreMap EP Mapping System.
Phase 2 Secondary Endpoints: | perioperatively/periprocedurally
  AF rhythm change or termination following CoreMap-guided ablation.
Phase 3 Secondary Endpoints: | perioperatively/periprocedurally
  AF rhythm change or termination following CoreMap-guided ablation vs. PVI+PW ablation of control arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Praha Klanovice, Czechia

IPD SHARING:
Plan to Share IPD: No